CLINICAL TRIAL: NCT02109757
Title: Evaluation of Hearing Protection Fit Testing Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Quintin Hecht, Hearing Conservation Program Manager, Doctor of Audiology, United States Air Force
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FWR20130114H
Record Dates: First submitted 2014-01-09; First posted 2014-04-10 (Estimated); Last update posted 2014-04-10 (Estimated); Status verified 2014-04

CONDITIONS: Hearing Loss
Keywords: Hearing conservation; Personal attenuation rating; earplug
MeSH Terms: conditions — Hearing Loss | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Software intervention and education (Experimental): This group will receive software intervention and education before and after receiving one-on-one education, thus showing if benefit or effect occurs simply due to having the software input before receiving education.
  Interventions: Other: Software intervention and education
- Education only (Active Comparator): This group will not receive software intervention prior to and after one-on-one education, only afterwards.
  Interventions: Other: Education only

INTERVENTIONS:
Other: Software intervention and education — Personal attenuation rating measurements will be taken before and after educating the patient using software program
  Arms: Software intervention and education
Other: Education only
  Arms: Education only

SUMMARY:
The specific aim of this research is to evaluate the performance, effectiveness, and long-term training benefits of a formal hearing protection fit testing program. This study may provide preliminary evidence on the benefits of direct education/training combined with a formal hearing protection device (HPD) fit testing on HPD fittings on United States Air Force (USAF) employees. Currently, Public Health provides informal, subjective training to employees; this practice may be altered by the results of this study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be enrolled in the hearing conservation program, and can be civilian or active duty/uniformed. Subjects must be currently using some form of in-the-ear hearing protection device on a regular basis and have ear canals free of cerumen, infection, or any other obstruction.

Exclusion Criteria:

* Not enrolled in the hearing conservation program. Not using in-the-ear hearing protection device on a regular basis. Ear canals containing cerumen, infection, or other obstructions.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Degree of earplug fit for participants in the Air Force Hearing Conservation Program as a measure of education and personnal attenuation rating. | 6 mos after intial subject visit
  The experimental group will show an increase, larger than the control group, in the amount of personal attenuation rating measurement shown by the software program as a result of software intervention used before and after education at the initial and follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Quintin A Hecht, Au.D., Principal Investigator — United States Air Force School of Aerospace Medicine
Locations (2):
- United States (2):
  - Elmendorf Air Force Base, Elemendorf Air Force Base, Alaska
  - Wright-Patterson Air Force Base, Dayton, Ohio